CLINICAL TRIAL: NCT06132256
Title: A 26-Week, Randomized, Double-Blind, Placebo-Controlled, Multi-center Study to Evaluate the Efficacy, Safety, and Tolerability of Axatilimab in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: MAXPIRe: Study to Evaluate Axatilimab in Participants With Idiopathic Pulmonary Fibrosis (IPF)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Collaborators: DevPro Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNDX-6352-0506; 2022-502954-15-00 (Other: EU-CT)
Record Dates: First submitted 2023-11-09; First posted 2023-11-15 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — axatilimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Axatilimab (Experimental): Participants will receive axatilimab every 2 weeks during the 26-week Treatment Period.
  Interventions: Drug: Axatilimab
- Placebo (Placebo Comparator): Participants will receive placebo every 2 weeks during the 26-week Treatment Period.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Axatilimab — Administered as intravenous (IV) infusion
  Other Names: Niktimvo; SNDX-6352
  Arms: Axatilimab
Other: Placebo — Placebo to match axatilimab administered as IV infusion. Placebo will not contain active ingredient.
  Arms: Placebo

SUMMARY:
The study will evaluate the efficacy and safety of axatilimab in participants with IPF.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented diagnosis of IPF per the 2018 American Thoracic Society (ATS)/European Respiratory Society (ERS)/Japanese Respiratory Society (JRS)/Latin American Thoracic Society Clinical Practice Guideline (Raghu 2018).
* Chest high-resolution computed tomography (HRCT) performed within 12 months prior to first Screening Visit and according to the minimum requirements for IPF diagnosis by central review based on participant's HRCT only (if no lung biopsy is available) or based on both HRCT and lung biopsy (with application of the different criteria in either situation). If an evaluable HRCT <12 months prior to Screening is not available, an HRCT can be performed at first Screening Visit to determine eligibility, according to the same requirements as the historical HRCT. If a participant has an indeterminate usual interstitial pneumonia (UIP) pattern and their HRCT is >6 months old, if in the opinion of the Investigator their disease has progressed, an additional HRCT may be obtained and reviewed for eligibility.
* FVC ≥45% of predicted normal at Screening Visits.
* Forced expiratory volume in 1 second (FEV1)/FVC ≥0.7 at Screening Visits.
* DLco ≥30% and ≤90% of predicted, corrected for hemoglobin at first Screening Visit.

Key Exclusion Criteria:

* Abnormalities detected on electrocardiogram (ECG) of either rhythm or conduction that in the opinion of the Investigator are clinical significant. Participants with implantable cardiovascular devices (for example, pacemaker) affecting the QT interval time may be enrolled in the study based upon Investigator judgment following cardiologist consultation if deemed necessary, and only after discussion with the Medical Monitor.
* Emphysema present on ≥50% of the HRCT, or the extent of emphysema is greater than the extent of fibrosis, according to central review of the HRCT.
* Interstitial lung disease associated with known primary diseases (for example, connective tissue disease, sarcoidosis and amyloidosis), exposures (for example, radiation, silica, asbestos, and coal dust), or drugs (for example, amiodarone).
* Participants who cannot meet protocol-specified baseline stability criteria.
* Acute IPF exacerbation within 3 months prior to screening.
* Receiving nintedanib in combination with pirfenidone
* Receiving systemic corticosteroids equivalent to prednisone >10 milligrams (mg)/day or equivalent within 2 weeks prior to Screening.
* Use of any of the following therapies within 4 weeks prior to Screening and during the Screening Period, or planned during the study: imatinib, ambrisentan, azathioprine, mycophenolate mofetil, cyclophosphamide, cyclosporine A, tacrolimus, bosentan, methotrexate, inhaled treprostinil, phosphodiesterase-5 inhibitors, including sildenafil (unless for occasional use), prednisone at steady dose >10 mg/day or equivalent, or other investigational therapy.
* History of cigarette smoking or vaping within the previous 3 months.
* Female participant who is pregnant or breastfeeding.
* Previous exposure to study intervention or known allergy/sensitivity to study drug.
* Receiving an investigational treatment within 28 days of randomization.
* Inadequate IV access.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of decline in morning pre-dose trough forced vital capacity (FVC) (milliliter [mL]) | Baseline through Week 26

SECONDARY OUTCOMES:
Time to disease progression | Baseline through Week 26
  Disease progression is defined as absolute FVC percent predicted decline of ≥10%, or occurrence of lung transplant or all-cause death prior to Week 26.
Annualized rate of decline in FVC percent predicted over 26 weeks | Baseline through Week 26
Change in St. George's Respiratory Questionnaire (SGRQ) score from Baseline to Week 26 | Baseline, Week 26
Change in diffusion capacity for carbon monoxide (DLco % of predicted, corrected for hemoglobin) from Baseline to Week 26 | Baseline, Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Syndax Pharmaceuticals
Locations (82):
- Australia (9):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Wallace Street Specialist Centre, Brisbane, Queensland
  - Mater Misericordiae Ltd, South Brisbane, Queensland
  - Griffith University Clinical Trial Unit, Southport, Queensland
  - Mackay Hospital & Health Service, West Mackay, Queensland
  - Monash Health, Clayton, Victoria
  - St Vincent's Melbourne, Fitzroy, Victoria
  - Institute for Respiratory Health, Perth, Western Australia
- Belgium (2):
  - OLV Hospital Aalst, Aalst, Oost-Vlaanderen
  - AZ Groeninge, Kortrijk, West-Vlaanderen
- Canada (2):
  - Centre de Recherche Clinique - CHUS, Sherbrooke, Quebec
  - Dynamic Drug Advancement, Ajax
- Thomayer University Hospital, Prague, Czechia
- France (3):
  - Chu Brest, Brest
  - CHU Dijon, Dijon
  - CHU de Rennes, Rennes
- Germany (8):
  - Klinikum Konstanz, Innere Medizin, Pneumologie, Konstanz, Baden-Wurttemberg
  - Pneumologisches Studienzentrum München-West, Munich, Bavaria
  - Studienzentrum Dr. Claus Keller, Frankfurt am Main, Hessia
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Klinikum Chemnitz - Zentrum für klinische Studien, Chemnitz
  - Studienzentrum Dr. Keller, Frankfurt am Main
  - Asklepios Lungenklinik Gauting, Gauting
  - RoMed Klinikum Rosenheim, Rosenheim
- Italy (12):
  - Ospedale Colonnello D'Avanzo, Foggia, Apulia
  - GB Morgagni Hospital, Forlì, FC
  - ASST Santi Paolo e Carlo, Milan, Lombardy
  - San Gerardo, Monza, MB
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga, Torino, Orbassano
  - University of Padua, Padua, Padua
  - Azienda Ospedaliera Universitaria Senese, Siena, Tuscany
  - A.O.U. Policlinico "G. Rodolico - San Marco", Catania
  - Azienda Ospedaliero Universitaria di Careggi, Florence
  - AOU di Modena, Modena
  - AOU Città della Salute e della Scienza di Torino - Molinette, Molinette
  - ISMETT, Palermo
- Poland (4):
  - Vitamed Galaj I Cichomski sp.j., Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Mics Centrum Medyczne Bydgoszcz, Bydgoszcz
  - Makowskie Centrum medyczne Hamernia Sp zz, Maków Podhalański
  - Warmia and Mazury Center for Lung Diseases, Olsztyn
- Romania (3):
  - Clinica Lavinia Davidescu SRL, Oradea
  - University of Medicine and Pharmacy "Victor Babes" Timisoara Department of Pneumology, Timișoara
  - Clinical Hospital of Infectious Diseases and Pneumophysiology Dr.Victor Babeș Timișoara Department of Pneumology, Timișoara
- South Korea (11):
  - Inje University Haeundae Paik Hospital, Haeundae, Busan
  - Chonnam National University Hospital, Gwangju, Dong-gu
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul, Eunpyeong-gu
  - Konkuk University Medical Center, Seoul, Gwangjin-gu
  - Chung-Ang University Gwangmyeong Hospital, Gyeonggi-do, Gwangmyeong-si
  - Gachon University Gil Medical Center, Incheon, Namdong-gu
  - Asian Medical Center, Seoul, Songpa-gu
  - Jeonbuk National University Hospital, Jeonju
  - Korea University ANAM Hospital, Seoul
  - SoonChunHyang University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (16):
  - Hospital Universitario Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - University Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Puerta del Mar - Pneumology and Thoracic Surgery Department, Cadiz
  - Giromed Institute, Girona
  - Hospital Arnau de Vilanova, Lleida
  - Hospital Gregorio Marañon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Universitario Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville
- Taiwan (4):
  - E-Da Hospital, Kaohsiung City
  - Chang-Geng Medical Foundation Linkou Chang-Geng Memorial Hospital, Linkou District
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- United Kingdom (7):
  - Royal Papworth Hospital - Clincial Research Facility, Cambridge, Cambridgehsire
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Oxford University Hospitals NHS Trust, Oxford, Oxforshire
  - Gannochy Trust Clinical Research Suite, Perth, Scotland
  - Leeds Teaching Hospitals NHS Trust, Leeds, W York
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands
  - Hull University Teaching Hospitals NHS Trust (Castle Hill), Cottingham, YS

IPD SHARING:
Plan to Share IPD: No